CLINICAL TRIAL: NCT01817634
Title: ω3 Long-chain Polyunsaturated Fatty Acids for Healthy Growth and Development of Infants and Young Children in the Gilgel Gibe Hydroelectric Dam Area, Ethiopia.
Brief Title: ω3 LCPUFAs for Healthy Growth and Development of Infants and Young Children in Southwest Ethiopia
Acronym: OME³Jim
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Jimma University (Other); VLIR Institutional University Collaboration Programme (Unknown); Nutrition Tiers Monde (Unknown); Nutricia Research Fundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2012/334
Record Dates: First submitted 2013-03-20; First posted 2013-03-25 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Child Malnutrition
Keywords: Malnutrition.
MeSH Terms: conditions — Child Nutrition Disorders; Malnutrition | interventions — Corn Oil; Fish Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Food supplement Intervention - Capsule Intervention (Experimental): Omega 3 food supplement + Omega 3 capsule.
  Interventions: Dietary Supplement: Fish powder corn-soy blend'+ Fish oil capsule.
- Food Supplement Intervention - Capsule Control (Experimental): Omega 3 food supplement + Control Capsule.
  Interventions: Dietary Supplement: Fish powder corn-soy blend + corn oil capsule.
- Food Supplement Control - Capusle Intervention (Experimental): Food supplement control + Omega 3 Capsule.
  Interventions: Dietary Supplement: Corn-soy blend + fish oil capsule.
- Food Supplement Control - Capsule Control (Active Comparator): Food supplement control + Control Capsule.
  Interventions: Dietary Supplement: Corn-soy blend + corn oil capsule.

INTERVENTIONS:
Dietary Supplement: Fish powder corn-soy blend'+ Fish oil capsule. — Omega 3 food supplement: 500 mg DHA + EPA, daily for 12 months. Omega 3 capsule: 500 mg DHA + EPA, daily for 12 months.
  Arms: Food supplement Intervention - Capsule Intervention
Dietary Supplement: Fish powder corn-soy blend + corn oil capsule. — Omega 3 food supplement: 500 mg DHA + EPA, daily for 12 months. Control capsule: 0 mg DHA + EPA, daily for 12 months.
  Arms: Food Supplement Intervention - Capsule Control
Dietary Supplement: Corn-soy blend + fish oil capsule. — control food supplement: 0 mg DHA + EPA, daily for 12 months. Omega 3 capsule: 500 mg DHA + EPA, daily for 12 months.
  Arms: Food Supplement Control - Capusle Intervention
Dietary Supplement: Corn-soy blend + corn oil capsule. — control food supplement: 0 mg DHA + EPA, daily for 12 months. Control capsule: 0 mg DHA + EPA, daily for 12 months.
  Arms: Food Supplement Control - Capsule Control

SUMMARY:
New approaches are needed to prevent growth failure in children from low- and middle-income countries (LMIC). To date, nutrition intervention studies have focused on micronutrient and energy content of complementary foods and have yielded only small to moderate effects on growth and development. There appears to be a missing link that mediates and reduces the expected beneficial effect. Child populations in LMIC show an asymptomatic environmental enteropathy that is characterized by a reduced size of the small intestinal villi, decreased gut integrity and a chronic inflammatory response in the gut. Results from studies in industrialized countries suggest that ω3 long-chain polyunsaturated fatty acids (ω3 LCPUFAs) improve immune response and gut integrity. These reported beneficial effects could result in even more important physiological implications for children from LMIC and will ultimately contribute to their healthy growth and development.

The hypothesis of the OME³Jim study is that an increased intake of ω3 LCPUFAs through complementary foods and human milk has an effect on infant growth and development in a context of high malnutrition rates and low ω3 LCPUFAs intake. This study will identify whether intake by either or both mother and infant is more effective.

The specific objectives of the OME³Jim study are:

1. To test the effect of supplementing infants with an ω3 LCPUFAs fortified food supplement on infant growth, morbidity, nutritional status and development;
2. To test the effect of supplementing lactating mothers with an ω3 LCPUFAs oil capsule on infant growth, nutritional status and development;
3. To test the combined effect (dose response) of supplementing ω3 LCPUFAs to lactating mothers and infant on infant growth, morbidity, nutritional status and development:
4. To test the effect of ω3 LCPUFAs supplementation on ω3 LCPUFA status in infants and human milk.

ELIGIBILITY:
Inclusion Criteria:

* Singleton infants
* 6-12 months old
* Not suffering from acute malnutrition (wasting): WHZ > -2 , no edema
* Infants currently being breastfed
* Anticipated local residence for the study duration
* Not planning to leave the study area for more than 1 month

Exclusion Criteria:

* Current supplement use or medical treatment of infant and/or mother
* Infants developing severe anemia (<70 g/L) or edema are referred to the nearby health institution for evaluation and treatment, and are omitted from the trial
* Presence of congenital abnormalities

Ages: 6 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 720 (Actual)
Dates: Start 2013-11; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in length-for-age Z-score over time up to 12 months. | Every month since baseline until 12 months.
  Length-for-age Z-score using the WHO 2006 growth reference chart.
Development score after study inclusion until 12 months after inclusion. | 6-monthly since baseline up to 12 months.
  Development score: Denver II test and Ages-Stages Social-Emotional Questionnaire.

SECONDARY OUTCOMES:
Weight-for-length Z-score up to 12 months. | 6-monthly up to 12 months.
  Weight-for-length Z-score: WHO 2006 growth reference chart.
Head circumference up to 12 months after inclusion | Monthly up to 12 months after inclusion
  Head circumference measurement.
Mid-upper arm circumference up to 12 months after inclusion. | Monthly until 12 months after inclusion.
  Mid-upper arm circumference.
Prevalence of stunting (HAZ <-2- up to 12 months after inclusion. | 6-monthly until 12 months after inclusion.
  According to WHO 2006 growth reference chart.
Prevalence of wasting (WHZ <-2) until 12 months after inclusion. | 6-monthly until 12 months after inclusion
  According to WHO 2006 growth reference chart.
C-reactive protein concentration until 12 months after inclusion | 6-monthly until 12 months after inclusion
  C-reactive protein concentration.
Haemoglobin concentration until 12 months | 6-monthly until 12 months after inclusion
  Haemoglobin concentration in blood sample.
Infant morbidity at weekly intervals. | weekly until 12 months after inclusion
  Infant morbidity (acute respiratory infection, diarrhoea, fever, malaria): weekly recall by caregiver, malaria by microscopy.
Breast milk concentrations of DHA/EPA/AA until 12 months after inclusion | 6-monthly until 12 months after inclusion
  Breast milk collections to determine milk levels of DHA/EPA/AA.
Infant blood concentrations of DHA/EPA/AA until 12 months after inclusion. | 6-monthly until 12 months after inclusion
  Blood sample for measuring infant blood levers of DHA/EPA/AA.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Kolsteren, MD, PhD, Principal Investigator — University Ghent
Locations (1):
- Jimma University, Jimma, Ethiopia

REFERENCES:
- [Derived] Argaw A, Bouckaert KP, Wondafrash M, Kolsteren P, Lachat C, De Meulenaer B, Hanley-Cook G, Huybregts L. Effect of fish-oil supplementation on breastmilk long-chain polyunsaturated fatty acid concentration: a randomized controlled trial in rural Ethiopia. Eur J Clin Nutr. 2021 May;75(5):809-816. doi: 10.1038/s41430-020-00798-x. Epub 2020 Nov 6. PMID 33159163
- [Derived] Argaw A, Huybregts L, Wondafrash M, Kolsteren P, Belachew T, Worku BN, Abessa TG, Bouckaert KP. Neither n-3 Long-Chain PUFA Supplementation of Mothers through Lactation nor of Offspring in a Complementary Food Affects Child Overall or Social-Emotional Development: A 2 x 2 Factorial Randomized Controlled Trial in Rural Ethiopia. J Nutr. 2019 Mar 1;149(3):505-512. doi: 10.1093/jn/nxy202. PMID 30544211
- [Derived] Argaw A, Wondafrash M, Bouckaert KP, Kolsteren P, Lachat C, Belachew T, De Meulenaer B, Huybregts L. Effects of n-3 long-chain PUFA supplementation to lactating mothers and their breastfed children on child growth and morbidity: a 2 x 2 factorial randomized controlled trial in rural Ethiopia. Am J Clin Nutr. 2018 Mar 1;107(3):454-464. doi: 10.1093/ajcn/nqx057. PMID 29566189